CLINICAL TRIAL: NCT04367935
Title: Effect of Pentoxifylline on Endothelial Dysfunction in Patients With Acute Coronary Syndrome: A Pilot Study
Brief Title: Effect of Pentoxifylline on Endothelial Dysfunction in Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Asmaa Saeed Mohamed Monir, Teaching Assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHCL 289
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Pentoxifylline; Endothelial Dysfunction; Oxidative Stress
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Pentoxifylline tablets 400mg three times daily for 2 months
  Interventions: Drug: Pentoxifylline
- Control (No Intervention): Control Group receiving placebo tablets three times daily for 2 months

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline tablets 400mg three times daily for 2 months
  Arms: Intervention

SUMMARY:
This study aims to investigate the effect of pentoxifylline administration on the status of endothelial function and oxidative stress biomarkers in patients with Acute Coronary Syndrome (ACS).

DETAILED DESCRIPTION:
The study will be carried out at Ain Shams University Hospitals. Patients with ACS who meet the eligibility criteria and consent to participate in the study will be randomly allocated to either the intervention group or the control group.

All participants will receive the standard pharmacologic treatment for ACS according to the applied guidelines offered by the facility. In addition, patients in the intervention group will receive Pentoxifylline tablets 400mg orally three times daily.

Patient follow-up will be scheduled every 2 weeks for each patient to check the tolerability, the development of side effects, any medication change and medication adherence. Physical examination at each visit will be done by physician in attendance for all patients in both groups.

A blood sample will be taken at baseline and at the end of the study after 2 months. for measurement of basic laboratory parameters (Complete Blood Count, Liver Function Tests, Kidney Function Tests ,..etc), the level of Soluble Vascular Cell Adhesion Molecule-1 (sVCAM-1) as a marker for endothelial dysfunction, the level of Malondialdehyde (MDA) as a marker for oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old.
* Recent ACS diagnosed-patients within the past 2 weeks.

Exclusion Criteria:

* Known allergy to pentoxifylline
* Heart failure New York Heart Association (NYHA) class III or IV
* Severe Left Ventricular Dysfunction (left ventricular ejection fraction <30%)
* High Serum creatinine level ≥ 2 mg/dl
* Liver disease (baseline alanine transaminase >2.5 times the upper limit of normal)
* Active bleeding or bleeding diathesis
* Major surgery or trauma within 1 month
* Recent cerebral and/or retinal hemorrhage within 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Level of Soluble Vascular Cell Adhesion Molecule-1 (sVCAM-1) as a marker for endothelial dysfunction | Two months
  will be measured at baseline and after 2 months

SECONDARY OUTCOMES:
Level of Malondialdehyde (MDA) as a marker for oxidative stress | Two months
  will be measured at baseline and after 2 months
Occurrence of side effects and Major Adverse Cardiac Events (MACE) | Two Months
  recorded rate of occurrence in both groups at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Saeed, Bachelor, Principal Investigator — Teaching Assistant at the Faculty of Pharmacy, Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Saeed A, Farouk MM, Sabri NA, Saleh MA, Ahmed MA. Effect of pentoxifylline on endothelial dysfunction, oxidative stress and inflammatory markers in STEMI patients. Future Sci OA. 2024 May 15;10(1):FSO967. doi: 10.2144/fsoa-2023-0266. eCollection 2024. PMID 38817362